CLINICAL TRIAL: NCT05778864
Title: Pharmacokinetics of LY3473329 Following Oral Administration in Participants With Renal Impairment Compared With Participants With Normal Renal Function
Brief Title: A Study of LY3473329 in Participants With Impaired and Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18638; J2O-MC-EKBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY3473329 (Control) (Experimental): LY3473329 administered orally to participants with normal renal function
  Interventions: Drug: LY3473329
- LY3473329 (Mild Renal Impairment) (Experimental): LY3473329 administered orally to participants with mild renal impairment
  Interventions: Drug: LY3473329
- LY3473329 (Moderate Renal Impairment) (Experimental): LY3473329 administered orally to participants with moderate renal impairment
  Interventions: Drug: LY3473329
- LY3473329 (Severe Renal Impairment) (Experimental): LY3473329 administered orally to participants with severe renal impairment
  Interventions: Drug: LY3473329
- LY3473329 (End-Stage Renal Disease) (Experimental): LY3473329 administered orally to participants with end-stage renal disease
  Interventions: Drug: LY3473329

INTERVENTIONS:
Drug: LY3473329 — Administered orally.

SUMMARY:
The main purpose of this study is to assess the amount of study drug (LY3473329) that reaches the bloodstream and the time it takes for the body to get rid of it when given to participants with renal (kidney) impairment compared to participants with normal renal function. The safety and tolerability of LY3473329 will also be evaluated in these participants. The study will last up to 8 weeks including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index within the range 19.0 to 42.0 kilograms per meter squared (kg/m²)
* Men who agree to use highly effective or effective methods of contraception, women of childbearing potential (WOCP) who agree to use highly effective or effective methods of contraception, and women not of childbearing potential (WNOCBP) may participate in this trial
* Have clinical laboratory test results within the normal reference range for the population

Exclusion Criteria:

* Have a history or presence of an underlying disease, or surgical, physical, medical, or psychiatric condition that, in the opinion of the investigator, would potentially affect participant safety within the study
* Have any abnormality in the 12-lead electrocardiogram (ECG), blood pressure and/or pulse rate that, in the opinion of the investigator, increases the risks associated with participating in the study
* Hemoglobin less than 8 grams/deciliter (g/dL) and/or clinically significant anemia symptoms
* Have an average weekly alcohol intake that exceeds 21 units per week for males and 14 units per week for females or males older than 65 years of age
* Smoke more than 10 cigarettes per day or the equivalent
* Have donated blood of more than 500 milliliter (mL) within 3 months prior to screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve from time zero to infinity (AUC0-∞) of LY3473329 | Predose up to 34 days postdose
  PK: AUC0-∞ of LY3473329
PK: Area under the concentration versus time curve from time zero to last time point (AUC0-tlast) of LY3473329 | Predose up to 34 days postdose
  PK: AUC0-tlast of LY3473329
PK: Maximum observed concentration (Cmax) of LY3473329 | Predose up to 34 days postdose
  PK: Cmax of LY3473329

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No